CLINICAL TRIAL: NCT04674475
Title: OPTImized Coronary Interventions eXplaIn the bEst cliNical outcomEs
Acronym: OPTI-XIENCE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Raul Moreno, MD, PhD, Director of Interventional Cardiology, Hospital La Paz, Madrid, Spain, Spanish Society of Cardiology
Other Study IDs: SpanishSC
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pressure guidewire, optimal coherence tomography — Pressure guidewire, optimal coherence tomography

SUMMARY:
Hypothesis: the clinical outcome of patients with indication of PCI and coronary stent implantation that are at high risk of events can be improved with a widespread use of intra-coronary tools that allow a PCI optimization (i.e. functional assessment by pressure guidewire and intra-coronary imaging techniques).

Objective: to evaluate whether the use of pressure guidewire and intra-coronary imaging techniques (mainly optimal coherence tomography) in patients at high risk of events undergoing coronary angiography for myocardial revascularization is associated with an improved clinical outcome in comparison with patient with angiographic alone guided cobalt-chromium everolimus-eluting coronary stenting.

Methods: Prospective observational multicentric international study with a follow-up of 12 months, including 1.000 patients in 40 sites located in 3 European countries (Spain, France, and Portugal). The control group will be comprised by a similar number of matched patients included in the "extended-risk" cohort of the XIENCE V USA study. PCI will be performed following local standard protocols and accordingly to the physician criteria. The use of pressure guidewire will be recommended according to the current guidelines, in patients with angiographically intermediate lesions and in those with multivessel disease. The use of OCT will be strongly recommended, as patients included will be considered to be at high risk of events, accordingly to the current recommendations. The primary endpoint will be target lesion failure (TLF) at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* At least one of the following high-risk characteristics: lesion length > 28 mm; reference vessel diameter < 2.5 mm or > 4.25 mm; chronic total occlusion; bifurcation with side branch ≥ 2 mm; ostial lesion; left main; in-stent restenosis; more than 2 lesions stented in the save vessel; more than 2 vessels treated; acute myocardial infarction; renal insufficiency; ejection fraction < 30%; or staged procedure. There will be no protocol exclusions on the basis of clinical features or angiographic criteria. The indication of using CCEES will be determined by the implanting physician.
* Informed consent signed

Exclusion Criteria:

* Patients whose survival is expected to be lower than 1 year at hospital discharge.
* Patients not willing to participate
* Patient not simultaneously participating in any interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective observational multicentric international study with a follow-up of 12 months, including 1.000 patients treated with coblat-chromium everolimus-eluting coronary stents and high risk of events in 40 sites located in 3 European countries (Spain, France, and Portugal). The control group will be comprised by a similar number of matched patients included in the "extended-risk" cohort of the XIENCE V USA study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-03 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-06-16 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 1 year
  composite of ischemia-driven target lesion revascularization, myocardial infarction (MI) related to the target vessel, or cardiac death related to the target vessel.

IPD SHARING:
Plan to Share IPD: Undecided